CLINICAL TRIAL: NCT00595465
Title: Comparison of Three Commercial Batches of the Japanese Encephalitis Vaccine IC51. Double Blind, Randomized, Controlled Phase 3 Study.
Brief Title: Comparison of Three Commercial Batches of the Japanese Encephalitis Vaccine IC51
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IC51-310
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Results first posted 2012-11-20 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- IC51 Batch A (Active Comparator)
  Interventions: Biological: Japanese Encephalitis purified inactivated vaccine
- IC51 Batch B (Active Comparator)
  Interventions: Biological: Japanese Encephalitis purified inactivated vaccine
- IC51 Batch C (Active Comparator)
  Interventions: Biological: Japanese Encephalitis purified inactivated vaccine

INTERVENTIONS:
Biological: Japanese Encephalitis purified inactivated vaccine — IC51 6 mcg i.m. injection on Day 0 and Day 28

SUMMARY:
The objective is to demonstrate equivalence of three commercial IC51 batches in terms of geometric mean titers for anti-JEV neutralizing antibody

ELIGIBILITY:
Main Inclusion Criteria:

* Male and female healthy adults aged at least 18 years, with written informed consent and either no childbearing potential or negative pregnancy test

Main Exclusion Criteria:

* History of immunodeficiency or immunosuppressive therapy,
* Known Human Immunodeficiency Virus (HIV); OR
* Drug addiction including alcohol dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Haas, Study Director — Valneva Austria GmbH
Locations (4):
- Medizinische Universität Wien, Universitätsklinik für Klinische Pharmakologie, Vienna, Austria
- Germany (3):
  - Berliner Zentrum Reise- und Tropenmedizin, Berlin
  - Klinikum der Universität München, Abteilung für Infektions- und Tropenmedizin, Munich
  - Klinik und Poliklinik für Innere Medizin der Universität Rostock, Rostock

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IC51 Batch IC51/07E/006A | IC51 Batch IC51/07E/007A | IC51 Batch IC51/07E/008A
Started | 130 | 129 | 128
Completed | 124 | 125 | 121
Not Completed | 6 | 4 | 7
Not completed — Adverse Event | 4 | 3 | 3
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — administrative reason | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IC51 Batch IC51/07E/006A | IC51 Batch IC51/07E/007A | IC51 Batch IC51/07E/008A | Total
Number analyzed (Participants) | 130 | 129 | 128 | 387
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 130 | 128 | 127 | 385
  >=65 years | 0 | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (8.6) | 28.9 (9.4) | 30.2 (10.5) | 29.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 83 | 74 | 228
  Male | 59 | 46 | 54 | 159
Region of Enrollment [Number; unit: participants]
  Europe | 130 | 129 | 128 | 387

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) for Anti-JEV Neutralizing Antibody
Time Frame: Day 56
Population: Per Protocol Population (PP Population, N= 364): includes all subjects randomized who received at least one dose of study medication without any major protocol violations identified at the blind data review meeting.
Measure: Mean (Standard Deviation); unit: titers
Arm/Group | IC51 Batch IC51/07E/006A | IC51 Batch IC51/07E/007A | IC51 Batch IC51/07E/008A
Number analyzed (Participants) | 124 | 121 | 119
titers | 160.8 (398.0) | 188.2 (410.2) | 168.4 (483.6)

2. Secondary Outcome: Seroconversion Rate
Time Frame: Day 56
Reporting Status: Not Posted

3. Secondary Outcome: Safety and Adverse Events
Time Frame: Day 56
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: 389 subjects were randomized, 2 of them were not treated
Arm/Group | IC51 Batch IC51/07E/006A | IC51 Batch IC51/07E/007A | IC51 Batch IC51/07E/008A
Serious Adverse Events (participants affected / at risk) | 2/130 | 1/129 | 0/128
Other Adverse Events (participants affected / at risk) | 64/130 | 74/129 | 74/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IC51 Batch IC51/07E/006A (N=130) | IC51 Batch IC51/07E/007A (N=129) | IC51 Batch IC51/07E/008A (N=128)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Tubo-Ovarian Abscess (Infections and infestations) | 1 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IC51 Batch IC51/07E/006A (N=130) | IC51 Batch IC51/07E/007A (N=129) | IC51 Batch IC51/07E/008A (N=128)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 4 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 3
Nausea (Gastrointestinal disorders) | 12 | 10 | 9
Vomiting (Gastrointestinal disorders) | 2 | 3 | 4
Fatigue (General disorders) | 17 | 19 | 14
Influenza Like Illness (General disorders) | 19 | 25 | 25
Injection Site Haematoma (General disorders) | 2 | 4 | 2
Injection Site Pain (General disorders) | 4 | 5 | 1
Pyrexia (General disorders) | 8 | 3 | 3
Bronchitis (Infections and infestations) | 3 | 4 | 2
Gastroenteritis (Infections and infestations) | 1 | 2 | 3
Nasopharyngitis (Infections and infestations) | 7 | 9 | 7
Rhinitis (Infections and infestations) | 3 | 3 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 10 | 15
Headache (Nervous system disorders) | 23 | 36 | 38
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other